CLINICAL TRIAL: NCT00768846
Title: Randomized Comparison of Zotarolimus- and Everolimus-Eluting Stents for Coronary Treatment
Brief Title: Zotarolimus and Everolimus-Eluting Stents ProsPectively Compared in Real World
Acronym: ZEPPELIN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Prof. Dr. A. Schoemig, Klinik fuer Herz- und Kreislauferkrankungen, Deutsches Herzzentrum Muenchen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. S03008
Record Dates: First submitted 2008-10-06; First posted 2008-10-08 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Coronary Artery Disease
Keywords: PCI; Stent; DES; CAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Endeavor Resolute Stent
  Interventions: Device: Endeavor Resolute Stent
- 2 (Active Comparator): Xience V Stent
  Interventions: Device: Xience V Stent

INTERVENTIONS:
Device: Endeavor Resolute Stent — Zotarolimus-eluting Endeavor Resolute Stent
  Arms: 1
Device: Xience V Stent — Everolimus-eluting Xience V Stent
  Arms: 2

SUMMARY:
The zotarolimus-eluting Endeavor Resolute stent is not inferior to the everolimus- eluting Xience V stent platform regarding a composite of cardiac death, myocardial infarction or target lesion revascularisation in a real-world population.

DETAILED DESCRIPTION:
The use of stents has become common practice in the percutaneous treatment of coronary artery disease. Restenosis affected 20-40% of de novo coronary lesions treated with bare metal stents. Drug-eluting stents (DES) have emerged as the most effective strategy for the prevention of restenosis. The first available DES were the Sirolimus-eluting Cypher and the Paclitaxel-eluting Taxus stent. Although their mid-term efficacy has been well-established, there is an ongoing debate on the potential of an increased incidence of late stent thrombosis, as well as of delayed onset of restenosis or catch-up phenomenon with DES. Recent evidence demonstrates that there might be differences between various DES in terms of safety and efficacy. The differences might be related to the drug, polymer or stent design. Everolimus (SDZ-RAD) and zotarolimus (ABT-578) are new antiproliferative agents that share some common structural and biological properties with sirolimus ("limus-group"). Both drugs bind to the intracellular sirolimus receptor, FK 506-binding protein 12 (FKBP 12). The drug-FKBP12 complex inhibits cell cycle progression via inactivation of the mammalian target of Rapamycin (mTOR) thereby regulating vascular smooth muscle cell migration and proliferation. Preclinical studies showed improved endothelialization and limited chronic inflammation of the everolimus-eluting stent compared with previous drug-eluting stents. Moreover, first randomized clinical trials of everolimus-eluting stents have shown promising results regarding safety, feasibility and efficacy in the suppression of neointimal proliferation. Safety and efficacy of the zotarolimus-eluting Endeavor stent have been investigated in the Endeavor clinical program. In the Endeavor III and IV trials, the Endeavour stent proved inferior to the Cypher and Taxus stents regarding angiographic endpoints. However, rates of target vessel failure were similar in both groups. The Endeavor RESOLUTE stent platform uses a new polymer with potential improvements of drug release compared to the Endeavor stent. The RESOLUTE clinical trial is the first-in man, observational, uncontrolled, non-randomized study evaluating the Endeavor Resolute drug-eluting stent with the new polymer. The trial enrolled a total of 130 patients with native coronary artery lesions. There are no data available comparing the zotarolimus-eluting Endeavor Resolute stent with the everolimus-eluting Xience V stent. Thus the aim of this prospective, randomized study is to compare the efficacy and safety of these two "new generation" drug-eluting stent platforms in a real world population.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years with symptomatic coronary artery disease undergoing PCI with stent implantation.
* Written, informed consent by the patient or her/his legally-authorized representative for participation in the study.

Exclusion Criteria:

* Cardiogenic shock.
* Malignancies or other comorbid conditions (for example severe liver, renal and pancreatic disease) with life expectancy less than 12 months or that may result in protocol non-compliance.
* Known allergy to the study medications: everolimus, zotarolimus, cobalt chrome.
* Inability to take clopidogrel for at least 6 months.
* Pregnancy (present, suspected or planned) or positive pregnancy test. (In women with childbearing potential a pregnancy test is mandatory.)
* Previous enrollment in this trial.
* Patient's inability to fully cooperate with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2600 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-05 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
A composite of cardiac death, myocardial infarction related to the target vessel or target lesion revascularisation | 1 year after randomization

SECONDARY OUTCOMES:
Late luminal loss | 6-8 months
Binary angiographic restenosis | 6-8 months
All cause mortality | 1 year
Stent thrombosis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Kastrati, MD, Study Chair — Deutsches Herzzentrum Munich; Julinda Mehilli, MD, Principal Investigator — Deutsches Herzzentrum Munich
Locations (2):
- Germany (2):
  - 1st Medizinische Klinik Klinikum rechts der Isar, Munich
  - Deutsches Herzzentrum Munich, Munich